CLINICAL TRIAL: NCT06600555
Title: CHANGE Evaluation of the Metabolic Surgery Technique for Glycemic Improvement in Type 2 Diabetes
Brief Title: Evaluation of the Metabolic Surgery Technique for Glycemic Improvement in Type 2 Diabetes
Acronym: CHANGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Médipôle Lyon-Villeurbanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHANGE metabolic surgery
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metabolic surgery with SLEEVE technique (Experimental)
  Interventions: Procedure: metabolic surgery with SLEEVE technique
- metabolic surgery with BY-PASS technique (Experimental)
  Interventions: Procedure: metabolic surgery with BY-PASS technique

INTERVENTIONS:
Procedure: metabolic surgery with SLEEVE technique — metabolic surgery with SLEEVE technique
  Arms: metabolic surgery with SLEEVE technique
Procedure: metabolic surgery with BY-PASS technique — metabolic surgery with BY-PASS technique
  Arms: metabolic surgery with BY-PASS technique

SUMMARY:
Surgery is one of the management options for type 2 diabetes in patients with moderate obesity. This is a recent option because it has been part of the recommendations since October 2022.

The possible surgical techniques are the same as those for bariatric surgery:

* Sleeve,
* Bypass,
* Gastric band, but the main goal is not weight loss, it is remission of type 2 diabetes. It is called metabolic surgery.

The ring technique (gastroplasty) is practiced less and less in France because it is less effective in weight loss and is responsible for major discomfort.

Currently, metabolic surgery is one of the recommendations but no study has compared the effectiveness of the techniques with each other. One or other of the techniques can be chosen according to the preferences of the surgeon, the patient, the center, etc. but this choice is not made objectively, in the absence of comparative data.

This study would like to follow up on patients for whom metabolic surgery has been proposed by the doctor,.

If the surgery is accepted, this study would like to improve knowledge of the effectiveness of the different techniques, and thus demonstrate which metabolic surgery technique is preferred in terms of effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

* adult patient and ≤ 65 years old
* T2D patient, with individualized glycemic objectives not achieved, despite medical care, in particular diabetological and nutritional, also including adapted physical activity, well conducted according to current good practice recommendations, for at least twelve months
* BMI between 30 and 34.9 kg/m²
* patient well informed beforehand about metabolic surgery and the study
* multidisciplinary evaluation (including a diabetologist) and decision on medical treatment by CM (date prior to inclusion)
* medical assessment of an acceptable surgical risk
* patient affiliated to or beneficiary of a social security system
* patient having freely signed the written informed consent

Exclusion Criteria:

* severe cognitive or mental disorders
* severe and unstabilized eating behavior disorders
* dependence on alcohol and licit and illicit psychoactive substances
* illnesses endangering life in the short and medium term
* contraindications to general anesthesia
* absence of identified prior medical care and foreseeable inability of the patient to participate in lifelong medical monitoring
* history of bariatric surgery
* pregnant or breastfeeding woman, or having a very long-term pregnancy plan short term (< 2 years)
* adult patient under guardianship or curatorship
* patient deprived of liberty or under judicial decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2032-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
T2DM remission rate | 1 year after surgery
  HbA1c lower than 6.5% in the absence of antidiabetic treatment, partial, complete, prolonged remission or no remission between the 2 surgical techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Medipole Lyon Villeurbanne, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No